CLINICAL TRIAL: NCT01411956
Title: The Effect of a Targeted Video Intervention on Beliefs Regarding Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Academy of Family Physicians (Other)
Responsible Party: Jennifer L. Middleton, MD, MPH, FAAFP, University of Pittsburgh Department of Family Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: G0804
Record Dates: First submitted 2011-07-27; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Hypertension
Keywords: Health Behavior Theory; Patient Education; Hypertension; Health beliefs related to hypertension and hypertension treatment
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): This group viewed the intervention video, a 24-minute episode of the sitcom "White Coats," deliberately scripted with the five health behavior theory constructs we are testing.
  Interventions: Other: 24-minute video episode of patient education TV sitcom "White Coats"
- Control Group (Placebo Comparator): The control group viewed a 25-minute video on an unrelated subject (depression).
  Interventions: Other: Placebo video

INTERVENTIONS:
Other: 24-minute video episode of patient education TV sitcom "White Coats" — The series features a fictional married couple of Family Medicine physicians who work in the same practice, located in our community. In both their professional and private lives and, in moments both humorous and serious, these doctors teach patients about a wide variety of health topics. The intervention episode addressing hypertension will focus on three different patient-physician plot lines, which were developed to specifically address each of the beliefs about hypertension highlighted in the theoretical model (susceptibility, seriousness, barriers, self-efficacy and outcome efficacy.).
  Arms: Treatment Group
Other: Placebo video — The control group watched a 25-minute patient education video on depression.
  Arms: Control Group

SUMMARY:
Researchers have linked media messages such as television programs to multiple problematic health behaviors. The narrative style of many television programs-involving a plot, recurrent characters, entertaining situations, and familiar settings-makes them compelling and likely contributes to the powerful influence these programs can have on behavior. However, narrative messages are not frequently utilized for prosocial purposes. In particular, health education embedded in a narrative context has been neither commonly utilized nor carefully evaluated. Using constructs from two complementary theories of health behavior, family physicians in a large metropolitan region have developed a situation comedy entitled "White Coats" that aims to provide quality patient education. The program currently airs on a local public access channel. The objective of this project is to evaluate the effect of one particular episode of "White Coats" on patient beliefs regarding hypertension.

DETAILED DESCRIPTION:
1. Design Randomized, single-blinded controlled trial.
2. Participants/Setting Permission from our Institutional Review Board has already been granted for this project (IRB #PRO07020003), but we are in the process of reapplying based on our revisions in response to the JGAP's initial review (please see section Q below). Participants will be recruited from the patient population of our largest residency family health center. The family health center cares for a pool of approximately 5000 patients with low to moderate income. Its population is roughly 40% male and 60% female. The population is racially diverse (Caucasian=60%; African American=20%; Other=20%). In order to recruit our study sample, we will generate a random list of patients from this health center's electronic records. All selected individuals will be contacted to assess whether they meet study criteria. As listed in Appendix 2, only persons with a history of hypertension or risk factors for hypertension will be included. In this way, we will recruit 80 volunteers aged 18-65.
3. Procedure Selected individuals will participate in two sessions. The first will consist of the intervention with pre-testing and immediate post-intervention testing, and the second will consist of a follow-up survey two months after the intervention. We will offer a $15 incentive (local grocery store gift card) to participate at each of these two steps for a total incentive of $30. Study personnel will contact those patients identified in the random sample by telephone and will read them a complete recruitment form. Recruited subjects will make an appointment to meet the research assistant for the initial survey testing and intervention exposure. At this appointment, study personnel will obtain verbal assent. Participants will be randomized using block randomization, stratifying for gender and age, into control and treatment arms. The entire randomization scheme will be completed a priori. Subjects will not be informed of their status as either a control or intervention group participant (single-blinded).

   All subjects will be led to a private room and will be given 15 minutes to complete the pre-test (Appendix 3). Participants in the intervention group will watch a twenty-five minute episode of "White Coats." Participants in the control group will watch a twenty-five minute educational video about depression. Immediately following the interventions, all subjects will be administered post-tests (Appendix 4). The research assistant will contact participants two months later by telephone to schedule a time to return to the family health center to take the delayed post-test (Appendix 5).
4. Intervention The intervention will consist of a twenty-five minute episode of a local health education situation comedy television series. Two physicians affiliated with a Family Medicine Residency and Fellowship Program created and currently produce this television series, entitled "White Coats," which currently airs on a local cable public access channel. The series features a fictional married couple of Family Medicine physicians who work in the same practice, located in our community. In both their professional and private lives and, in moments both humorous and serious, these doctors teach patients about a wide variety of health topics. The intervention episode addressing hypertension will focus on three different patient-physician plot lines, which were developed to specifically address each of the beliefs about hypertension highlighted in the theoretical model (susceptibility, seriousness, etc.).
5. Measures Evaluation will consist of pre- and post-testing, both immediate and at a two-month follow-up, with a self-administered written survey. The primary outcome measures will consist of five items (Q15-Q19) representing constructs from the health belief model and social cognitive theory: (1) perceived seriousness of hypertension (Q15), (2) perceived susceptibility to hypertension (Q16), (3) barriers to hypertension control (Q17), (4) self-efficacy regarding hypertension control (Q18), and (5) outcome efficacy regarding hypertension control (Q19). All outcomes will be scored on a 1 to 7 point Likert scale. We have modeled question items from existing reliable, valid instruments,23-25 although no complete previously validated instrument exists to specifically measure these five constructs as they relate to hypertensive control.

We will collect demographics including age as a continuous variable (based on date of birth), gender, race/ethnicity, and socioeconomic status. Race/ethnicity will be collected in the manner suggested by the National Institutes of Health, allowing participants to select more than one race/ethnicity. Socioeconomic status will be approximated with highest level of education achieved.

ELIGIBILITY:
Inclusion Criteria: age between 18 and 65, along with one or more of the following

* ever told by a physician that you have hypertension
* family history of hypertension
* current stress
* BMI over 30
* current smoker
* inactive/sedentary lifestyle (defined as less than 150 minutes of exercise a week)

Exclusion Criteria:

* age under 18 or over 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in Likert scale agreement with Perceived severity questionnaire statement from immediately pre-intervention to immediately post-intervention and also 2 months post-intervention | immediately pre-intervention, immediately post-intervention, and 2 months post-intervention
  Participants ranked their agreement with the following statement on an 8-point Likert scale: "If you have high blood pressure, controlling your blood pressure is important."
Change in Likert scale agreement with Perceived susceptibility questionnaire statement from immediately pre-intervention to immediately post-intervention and also 2 months post-intervention | immediately pre-intervention, immediately post-intervention, and 2 months post-intervention
  Participants ranked their agreement with the following statement on an 8-point Likert scale: "People don't need to worry about having high blood pressure if they don't have any symptoms (like headaches, chest pain, or blurry vision)."
Change in Likert scale agreement with Perceived barriers to change questionnaire statement from immediately pre-intervention to immediately post-intervention and also 2 months post-intervention | immediately pre-intervention, immediately post-intervention, and 2 months post-intervention
  Participants ranked their agreement with the following statement on an 8-point Likert scale: "I can find time to exercise."
Change in Likert scale agreement with self-efficacy questionnaire statement from immediately pre-intervention to immediately post-intervention and also 2 months post-intervention | immediately pre-intervention, immediately post-intervention, and 2 months post-intervention
  Participants ranked their agreement with the following statement on an 8-point Likert scale: "I can read food labels to look for high salt foods when I buy groceries."
Change in Likert scale agreement with Outcome efficacy questionnaire statement from immediately pre-intervention to immediately post-intervention and also 2 months post-intervention | immediately pre-intervention, immediately post-intervention, and 2 months post-intervention
  Participants ranked their agreement with the following statement on an 8-point Likert scale: "If you have high blood pressure and take your medicines, you can lower your chance of having a heart attack."

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Middleton, MD MPH FAAFP, Principal Investigator — University of Pittsburgh Department of Family Medicine